CLINICAL TRIAL: NCT05657951
Title: Repeatability and Reproducibility of Lens Zonule Length Measurement Using ArcScan Insight 100 Very High-frequency Digital Ultrasound
Brief Title: Repeatability and Reproducibility of Lens Zonule Length Measurement Using ArcScan Insight 100
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president, Wenzhou Medical University
Other Study IDs: Insight100-zonule1
Record Dates: First submitted 2022-11-29; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Zonule of Zinn Abnormality; Zonular Cataract
MeSH Terms: conditions — Cataract, zonular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal eyes
  Interventions: Device: ArcScan Insight 100 very high-frequency digital ultrasound

INTERVENTIONS:
Device: ArcScan Insight 100 very high-frequency digital ultrasound — The Insight-100 (ArcScan Inc., Golden, CO, USA) employs the high-frequency B-scan in the assessment of anterior segment parameters. Anormal saline coupling medium is formed with a disposable eyepiece between the 50 MHz transducer and the eye. The instrument moves the transducer in an arc so that the beam axis maintains approximate normality to the surface of the eye. The frequencies of cornea, anterior chamber, and lens are 60 MHz, 50 MHz and 50 MHz, respectively. The maximum arc scanning range is 70 degrees, and there is a linear scanning range of 29mm. The axial and lateral resolutions are 35 μm and 65 μm, respectively. It can measure structures behind the iris, including lens zonule.

SUMMARY:
The purpose of this study is to evaluate the intra-examiner repeatability and inter-examiner reproducibility in lens zonule length measurements using very high-frequency (VHF) digital ultrasound (ArcScan Insight 100).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with no ocular disease except ametropia
* Subjects will be able to understand and willing to sign an informed consent

Exclusion Criteria:

* Previous ocular surgery
* Subjects not being able to tolerate or not willing to use pilocarpine eye drops
* Subjects has active ocular infection or inflammation
* Subjects not being able to look steadily
* Subjects not being able to open eyes wide in sterile saline even after topical anesthesia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy subjects with no ocular disease except ametropia
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Repeatability of ArcScan Insight 100 zonule scans in normal eyes (standard deviation and coefficient of variation) | 1 day
  First, three images will be obtained under'capsule model'using ArcScan Insight 100, and the length of zonule will be measured with built-in software by operator A.
  Operator B then performed the measurements using the same procedure and technique.
  The standard deviation and coefficient of variation of 3 repeated measurements for zonule length. will be calculated.
Reproducibility of ArcScan Insight 100 zonule scans in normal eyes | 1 day
  First, three images will be obtained under'capsule model'using ArcScan Insight 100, and the length of zonule will be measured with built-in software by operator A.
  Operator B then performed the measurements using the same procedure and technique.
  The intraclass correlation is used to evaluate the difference between operator A and operator B.

SECONDARY OUTCOMES:
Repeatability of zonule length measurement with the built-in software (the intraclass correlation) | 1 month
  After a 1-month period, operator A and operator B will measure the zonule length again. The intraclass correlation is used to evaluate the difference between the two repeated measurements of one same image by Operator A or Operator B.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of WMU, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li X, Chang P, Li Z, Qian S, Zhu Z, Wang Q, Yun-E Z. Agreement between anterior segment parameters obtained by a new ultrasound biomicroscopy and a swept-source fourier-domain anterior segment optical coherence tomography. Expert Rev Med Devices. 2020 Dec;17(12):1333-1340. doi: 10.1080/17434440.2020.1848541. Epub 2020 Dec 1. PMID 33196325
- [Derived] Zhu Z, Zou H, Li H, Wu X, Wang Y, Li Z, Zhao Y. Repeatability and reproducibility of anterior lens zonule length measurement using ArcScan insight 100 very high-frequency ultrasound. Expert Rev Med Devices. 2023 Jul-Dec;20(8):703-710. doi: 10.1080/17434440.2023.2223967. Epub 2023 Jun 13. PMID 37300312